CLINICAL TRIAL: NCT03420937
Title: Deep Neuromuscular Block During General Anaesthesia in Laparoscopic (and Robotic Laparoscopic) Surgery and Its Potential Benefits for Certain Physiological Parameters in Perioperative Period
Brief Title: Deep Neuromuscular Block During General Anaesthesia in Robotic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, MUDr. Lenka Doubravska, MUDr. Lenka Doubravská, University Hospital Olomouc
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IGA_LF_2016_021
Record Dates: First submitted 2016-05-22; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Observation of Neuromuscular Block; Complication of Ventilation Therapy; Postoperative Recovery
Keywords: deep neuromuscular block; laparoscopic surgery; robotic surgery; lung protective ventilation; respiratory functions; post-operative recovery
MeSH Terms: interventions — Sugammadex; Neostigmine; Atropine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deep Neuromuscular Block (Experimental): Administration of rocuronium 0,6 mg/kg iv, top-ups 5-10 mg iv to target value of Post-tetanic Count (PTC) = 1-2; PTC measurement every 4 min.
  Intervention: Neuromuscular blockade reversal at the end of anesthesia: sugammadex 2 mg/kg iv (when PTC is 18-20 and TOF-count 0) or sugammadex 4 mg/kg iv (when PTC under 18).
  Induction of anesthesia: midazolam 1-2 mg iv, sufentanil 10-30 mcg iv, propofol 1,5-2,5 mg/kg iv Anesthesia: sevoflurane in air to target 1.2-1.5 minimal alveolar concentration (MAC). Rescue medication: sevoflurane, propofol 20-40 mg iv.
  Extubation when patient is conscious and attained recovery from neuromuscular blockade to a TOF-ratio of at least 0,9.
  Interventions: Drug: Sugammadex
- Moderate Neuromuscular Block (Experimental): Administration of rocuronium 0,6 mg/kg iv, top-ups 5-10 mg iv to target value of Train-of-Four (TOF) count = 1-2, TOF-count measurement every 1 min. Intervention: Neuromuscular blockade reversal at the end of anesthesia: neostigmine 0.03 mg/kg iv + atropine 0.5-1.0 mg iv Induction of anesthesia: midazolam 1-2 mg iv, sufentanil 10-30 mcg iv, propofol 1.5-2.5 mg/kg iv Anesthesia: sevoflurane in air to target 1.2-1.5 minimal alveolar concentration (MAC). Rescue medication: sevoflurane, propofol 20-40 mg iv Extubation when patient is conscious and attained the recovery from neuromuscular blockade to a TOF-ratio of at least 0,9.
  Interventions: Drug: Neostigmine, Atropin Biotika

INTERVENTIONS:
Drug: Sugammadex — Deep neuromuscular block provided by rocuronium to PTC 1-2. Reversal of the block with sugammadex.
  Other Names: Bridion
  Arms: Deep Neuromuscular Block
Drug: Neostigmine, Atropin Biotika — Standard neuromuscular block provided by rocuronium to TOF-count 1-2. Reversal of the block with neostigmine.
  Other Names: syntostigmine, atropine
  Arms: Moderate Neuromuscular Block

SUMMARY:
The aim of this project is to show, whether the use of the deep neuromuscular block in certain laparoscopic robot-assisted surgery can positively influence main physiological functions compared to the use of standard neuromuscular block. Secondary outcome is to find out whether the targeted specific reversal of neuromuscular block by sugammadex improves and fastens the post-operative recovery of the patients.

DETAILED DESCRIPTION:
Adequate muscle relaxation during general anaesthesia is crucial for easy, uncomplicated and safe laparoscopic and robot-assisted surgery. Perfect abdominal wall relaxation facilitates surgical working conditions, which makes surgery safer, faster and easier to perform. Besides this indirect advantage, there could be obvious benefit for patients. This is a result of decreased negative pathophysiological consequences of an increased intraabdominal pressure (capnoperitoneum) on important organ systems (cardiovascular, breathing system, kidneys etc.) Complete muscle relaxation during general anaesthesia can be achieved by using higher doses of rocuronium (non-depolarizing aminosteroid muscle relaxant) and special anaesthetic technique called deep neuromuscular block (DNMB). The primary focus of the project is to test the potential advantages of DNMB compared to standard relaxation technique. Safe and efficient use of NMBA is an important precondition in restoring a patient´s full muscle strength at the end of anaesthesia, to prevent effects of residual block. Modern practice of anaesthesia offers an option for complete and immediate rocuronium induced block reversal by using its specific antagonist - sugammadex. Combination of DNMB approach and sugammadex reversal also provide potential benefits for perioperative course and patient recovery after surgery. Secondary objective of the project is to verify this facts.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Informed Consent
* Elective robotic radical prostatectomy
* American Society of Anesthesiologists (ASA) status 1-3

Exclusion Criteria:

* Inability to obtain Informed ConsentAge under 18 years
* American Society of Anesthesiologists (ASA) status over 3
* Indication for rapid sequence induction, signs of difficult airway severe neuromuscular, liver or renal disease
* Known allergy to drugs used in the study
* Malignant hyperthermia (medical history)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Surgical conditions SRS | Perioperative period
  Describes the quality of surgical conditions as reported by surgeon
Intraabdominal pressure IAP (mmHg) | During surgery
  Pressure in the abdominal cavity during capnoperitoneum

SECONDARY OUTCOMES:
Operating theatre time (min) | during anesthesia
  Time from induction to anesthesia to the release from operating theatre
Post-operative recovery | post-operative period (1 week)
  Physiological functions, level of discomfort, subjective evaluation by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Karel Axmann, MD, Principal Investigator — University Hospital Olomouc
Locations (1):
- Dept. of Anesthesiology and Intensive Care Medicine, University Hospital Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs-Buder T, Claudius C, Skovgaard LT, Eriksson LI, Mirakhur RK, Viby-Mogensen J; 8th International Neuromuscular Meeting. Good clinical research practice in pharmacodynamic studies of neuromuscular blocking agents II: the Stockholm revision. Acta Anaesthesiol Scand. 2007 Aug;51(7):789-808. doi: 10.1111/j.1399-6576.2007.01352.x. PMID 17635389
- [Background] Blobner M, Frick CG, Stauble RB, Feussner H, Schaller SJ, Unterbuchner C, Lingg C, Geisler M, Fink H. Neuromuscular blockade improves surgical conditions (NISCO). Surg Endosc. 2015 Mar;29(3):627-36. doi: 10.1007/s00464-014-3711-7. Epub 2014 Aug 15. PMID 25125097
- [Background] Van Wijk RM, Watts RW, Ledowski T, Trochsler M, Moran JL, Arenas GW. Deep neuromuscular block reduces intra-abdominal pressure requirements during laparoscopic cholecystectomy: a prospective observational study. Acta Anaesthesiol Scand. 2015 Apr;59(4):434-40. doi: 10.1111/aas.12491. Epub 2015 Feb 13. PMID 25684372
- [Background] Madsen MV, Gatke MR, Springborg HH, Rosenberg J, Lund J, Istre O. Optimising abdominal space with deep neuromuscular blockade in gynaecologic laparoscopy--a randomised, blinded crossover study. Acta Anaesthesiol Scand. 2015 Apr;59(4):441-7. doi: 10.1111/aas.12493. Epub 2015 Mar 1. PMID 25789421
- [Background] Staehr-Rye AK, Rasmussen LS, Rosenberg J, Juul P, Lindekaer AL, Riber C, Gatke MR. Surgical space conditions during low-pressure laparoscopic cholecystectomy with deep versus moderate neuromuscular blockade: a randomized clinical study. Anesth Analg. 2014 Nov;119(5):1084-92. doi: 10.1213/ANE.0000000000000316. PMID 24977638
- [Background] Gerges FJ, Kanazi GE, Jabbour-Khoury SI. Anesthesia for laparoscopy: a review. J Clin Anesth. 2006 Feb;18(1):67-78. doi: 10.1016/j.jclinane.2005.01.013. PMID 16517337
- [Background] Gainsburg DM. Anesthetic concerns for robotic-assisted laparoscopic radical prostatectomy. Minerva Anestesiol. 2012 May;78(5):596-604. Epub 2012 Mar 13. PMID 22415437
- [Background] Carron M. Respiratory benefits of deep neuromuscular block during laparoscopic surgery in a patient with end-stage lung disease. Br J Anaesth. 2015 Jan;114(1):158-9. doi: 10.1093/bja/aeu419. No abstract available. PMID 25500396
- [Background] Kilpatrick B, Slinger P. Lung protective strategies in anaesthesia. Br J Anaesth. 2010 Dec;105 Suppl 1:i108-16. doi: 10.1093/bja/aeq299. PMID 21148650
- [Background] Futier E, Constantin JM, Jaber S. Protective lung ventilation in operating room: a systematic review. Minerva Anestesiol. 2014 Jun;80(6):726-35. Epub 2013 Nov 13. PMID 24226493
- [Background] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS. Residual neuromuscular blockade and critical respiratory events in the postanesthesia care unit. Anesth Analg. 2008 Jul;107(1):130-7. doi: 10.1213/ane.0b013e31816d1268. PMID 18635478
- [Background] Blobner M, Eriksson LI, Scholz J, Motsch J, Della Rocca G, Prins ME. Reversal of rocuronium-induced neuromuscular blockade with sugammadex compared with neostigmine during sevoflurane anaesthesia: results of a randomised, controlled trial. Eur J Anaesthesiol. 2010 Oct;27(10):874-81. doi: 10.1097/EJA.0b013e32833d56b7. PMID 20683334
- [Background] Rahe-Meyer N, Berger C, Wittmann M, Solomon C, Abels EA, Rietbergen H, Reuter DA. Recovery from prolonged deep rocuronium-induced neuromuscular blockade: A randomized comparison of sugammadex reversal with spontaneous recovery. Anaesthesist. 2015 Jul;64(7):506-12. doi: 10.1007/s00101-015-0048-0. Epub 2015 Jul 1. PMID 26126940
- [Background] Kopman AF, Naguib M. Laparoscopic surgery and muscle relaxants: is deep block helpful? Anesth Analg. 2015 Jan;120(1):51-58. doi: 10.1213/ANE.0000000000000471. PMID 25625254
- [Background] Carron M, Ori C. Deep Neuromuscular Blockade for Laparoscopy: A Different View. Anesth Analg. 2016 Jan;122(1):289. doi: 10.1213/ANE.0000000000000864. No abstract available. PMID 26678476
- [Result] Dubois PE, Putz L, Jamart J, Marotta ML, Gourdin M, Donnez O. Deep neuromuscular block improves surgical conditions during laparoscopic hysterectomy: a randomised controlled trial. Eur J Anaesthesiol. 2014 Aug;31(8):430-6. doi: 10.1097/EJA.0000000000000094. PMID 24809482